CLINICAL TRIAL: NCT04576390
Title: Palonosetron Versus Ondansetron for PONV Prevention in Patients Undergoing Endoscopic Retrograde Cholangio-Pancreatography ERCP: A Prospective Randomized Controlled Study
Brief Title: Palonosetron Versus Ondansetron for PONV Prevention in Patients Undergoing ERCP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Theodor Bilharz Research Institute (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Hanan Farouk Khafagy, Professor doctor, Theodor Bilharz Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TBRI -Palonosetron
Record Dates: First submitted 2020-09-23; First posted 2020-10-06 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-09

CONDITIONS: Antiemetic; Postoperative Nausea and Vomiting
Keywords: Palonosetron; Ondansetron; PONV; ERCP
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Ondansetron; Palonosetron

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group O (Active Comparator): On the day of procedure, the recruited patients in Group O will be given Ondansetron 4 mg diluted for up to 5ml using normal saline by a colleague not participating to the study or the patient care & will label the syringes as antiemetic.
  Interventions: Drug: Ondansetron 4 mg
- Group P (Active Comparator): On the day of procedure, the recruited patients in Group P will be given Palonosetron 75 mcg diluted for up to 5ml using normal saline by a colleague not participating to the study or the patient care & will label the syringes as antiemetic.
  Interventions: Drug: Palonosetron 75 mcg

INTERVENTIONS:
Drug: Ondansetron 4 mg — Antiemetic drug
  Other Names: Zofran
  Arms: Group O
Drug: Palonosetron 75 mcg — Antiemetic drug
  Other Names: Aloxi
  Arms: Group P

SUMMARY:
This study is designed to compare the effects of a single dose Ondansetron 4mg versus Palonosetron 75mcg in the prophylaxis against early & delayed postoperative nausea and vomiting in the first 48 hours post-operatively in patients undergoing Endoscopic Retrograde Cholangio-Pancreatography (ERCP) to determine the complete response, complete control and failure rates.

DETAILED DESCRIPTION:
Premedication will be omitted. Pre-operative baseline values of heart rate and blood pressure will be recorded. On arrival in the operation theatre, the routine monitoring devices (ECG, Pulse Oximetry & Non Invasive Blood Pressure) will be applied and base line heart rate, blood pressure (Systolic, diastolic and mean arterial blood pressure) and arterial Oxygen saturation will be recorded.

After an intravenous line is secured, while pre-oxygenating the patient. Anaesthesia will be induced using fentanyl 1-2 µg/kg and sodium propofol 1.5-2.5 mg/kg according to the patient general condition and hemodynamics and intubation will be facilitated by using atracurium besylate 0.5mg/kg.

Anaesthesia will be maintained with O2 in air (50%), sevoflurane (0.8-1.0 MAC). Muscle relaxation will be maintained with boluses of atracurium besylate 0.1 mg/kg. Intermittent positive pressure ventilation will be adjusted to maintain end tidal carbon dioxide between 30-35mm Hg. Intravenous crystalloids (3-4 ml/kg/hr) will infused during intra-operative and immediate post-operative period. Intra-operatively, the following parameters will be monitored: ECG, blood pressure, pulse rate, end tidal carbon dioxide (ET CO2) & oxygen saturation (SpO2). Diclofenac sodium 1mg/kg intramuscularly to protect against Post ERCP Pancreatitis & Paracetamol (1gm) intravenously will be administered 15 minutes before the end of procedure followed by the administration of the anti-emetic prophylaxis according to group allocation.

At the end, residual neuromuscular block will be antagonized using atropine and neostigmine and trachea will be extubated after signs of adequate neuro-muscular reversal are achieved. After extubation, patients will be transferred to the Post anaesthesia care unit where the blood pressure, heart rate, respiratory rate and O2 saturation will be monitored continuously every five minutes for 60 minutes.

If Visual Analogue Score (VAS) score is ≥3, rescue analgesia will be provided with Pethidine in 10mg increments / 5minutes until the VAS score is less than 3.

Pain intensity will be assessed using VAS for the first 24 hours. Post-operative pain relief will be provided Paracetamol (1gm) intravenously given regularly every 8 hours for the first 24 hours.

Any incidence of nausea, retching or vomiting and use of any rescue medication during the first 24 hours at time interval of 0, 1/2, 1, 2, 6,12, 24 and 48 h will be noted, Nausea is defined as the subjective sensation of an urge to vomit, in the absence of expulsive muscular movements. Retching is defined as an unproductive effort to vomit. Vomiting is defined as the forcible expulsion of the gastric contents through the mouth. Retching and vomiting will be collectively termed emetic episodes.

Rescue anti-emetic therapy in the form of Metoclopramide 10 mg intravenously will be provided for any patient suffering from an emetic episode as described above. The use of antiemetic rescue medication will be recorded & analysed.

Patients will stay at the hospital post ERCP according to the discretion of the treating physician opinion, if any patient will be discharged before 48 hours, the data will be collected by telephone.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-60 years of age
* American Society of Anaesthesiologists physical status (ASA) grade I-II
* 1 - 2 Risk factor for PONV according to Apfel Score

  o Apfel Score includes 4 points : Female gender, history of PONV and/or motion sickness, non-smoking status, and post-operative use of opioids , the risk of PONV is 10%, 20%, 40%,60% or 80% respectively
* Undergoing elective ERCP.
* Having provided written informed consent signed by patient or guardian.

Exclusion Criteria:

* Allergy to any drug being used in the study
* ASA III-IV
* History of vomiting, retching, nausea or antiemetics use in the 24 hours prior to day of procedure
* Patients receiving steroids, prokinetics, or antacids intake in the previous 48 hours
* Patients with significant gastro-oesophageal disease
* Menstruating, lactating or pregnant females
* History of alcohol or substance abuse
* Significant systemic disease of the liver, kidneys, heart, lungs, Cancer and or diabetes mellitus.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-10-24 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-05-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of PONV | During 24 hours post-operatively
  Incidence of nausea, retching or vomiting

SECONDARY OUTCOMES:
Incidence of PONV | During 48 hours post-operatively
  Incidence of nausea, retching or vomiting
Complete Responders | During 48 hours postoperatively
  Number of patients has no rescue medication and no emesis
Complete control | During 48 hours postoperatively
  Number of patients has no rescue medication, no emesis, no more than mild nausea
Failed prophylaxis | During 48 hours postoperatively
  Number of patients with episode of emesis and needs rescue medication
Time to rescue anti-emetics or emesis | Time in minutes during 48 hours postoperatively
  Time until patient takes antiemetic or emesis occurs

CONTACTS AND LOCATIONS:
Overall Officials: Omar M. Abou-Hashim, residant, Study Chair — Theodor Bilharz Research Institute; Yahia M. Hammad, Lecteurer, Study Director — Cairo University